CLINICAL TRIAL: NCT07070765
Title: Sodium-glucose Transporter Type 2 Inhibition in Anthracycline-related Cardiotoxicity - SPRINT
Brief Title: Sodium-glucose Transporter Type 2 Inhibition in Anthracycline-related Cardiotoxicity
Acronym: SPRINT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3-033-23
Record Dates: First submitted 2025-06-26; First posted 2025-07-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy; anthracycline; sodium-glucose transporter type 2 inhibition
MeSH Terms: conditions — Breast Neoplasms | interventions — Sodium-Glucose Transporter 2; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium-glucose transporter type 2 inhibition treatment arm (Active Comparator): Sodium-glucose transporter type 2 inhibition plus standard clinical care for the duration of chemotherapy treatment
  Interventions: Drug: Sodium-glucose transport-2 (SGLT-2) inhibitors
- Standard clinical care placebo treatment arm (Placebo Comparator): Standard clinical care for the duration of chemotherapy treatment
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: Sodium-glucose transport-2 (SGLT-2) inhibitors — Dapagliflozin 10mg in addition to standard clinical care
  Other Names: Dapagliflozin 10mg in addition to standard clinical care
  Arms: Sodium-glucose transporter type 2 inhibition treatment arm
Other: Standard medical treatment — Standard clinical care
  Other Names: Standard clinical care
  Arms: Standard clinical care placebo treatment arm

SUMMARY:
Cardiotoxicity is heart damage that arises from certain drugs, such as those used for cancer treatment and develops in approximately 10% of patients with breast cancer who are treated with anthracyclines. It has been suggested that sodium-glucose transporter-2 (SGLT2) inhibitors may reduce the damage to the heart caused by anthracycline chemotherapy. The investigators wish to determine whether dapagliflozin (SGLT2 inhibitor) taken daily during chemotherapy will reduce the rate of cardiotoxicity.

DETAILED DESCRIPTION:
Cardiac dysfunction is a major complication of cancer drug therapies, affecting approximately 10% of patients treated with anthracyclines. It has the worst prognosis of all cardiomyopathies and is currently thought to be a consequence of an energetic based mitochondrial dysfunction. This energy deficit could potentially be ameliorated by the putative cardiometabolic benefits of sodium-glucose transporter type 2 inhibition. In pilot data from patients with breast cancer, the investigators have demonstrated that cardiac magnetic resonance spectroscopy can identify and quantify the myocardial energetic deficit associated with anthracycline therapy. The purpose of this study is to determine whether sodium-glucose transporter type 2 inhibition has the potential to reverse the myocardial energetic deficit associated with anthracycline toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer between 18-70 years of age.
* Patients with low to medium cardiovascular risk.
* Patients scheduled for adjuvant or neo-adjuvant anthracycline therapy.
* Patients who are able to give written informed consent to take part in the study.
* Patients who can read and understand English.

The current thresholds for defining cardiovascular risk for patients undergoing anthracycline chemotherapy are as follows: normal resting 12-lead electrocardiogram, plasma cardiac troponin I concentration < 99th centile, serum brain natriuretic peptide concentration <35 pg/mL or serum N-terminal pro-brain natriuretic peptide concentration <125 pg/mL, left ventricular ejection fraction >55%, global longitudinal strain >-18% and healthy life-style (normal body-mass index, non-smoker). Low cardiovascular risk will allow for the presence of one abnormal life-style factor (body-mass index indicating obesity (>30 kg/m2), current smoker or significant smoking history), or presence of only one of the following in the clinical history: hypertension, stage 1-2 chronic kidney disease, age 65-79 years, borderline left ventricular ejection fraction (50-54%) or elevated cardiac biomarkers. Medium cardiovascular risk will permit the combination of any 2-4 of the lifestyle or clinical history variables indicated above.

Exclusion Criteria:

* Patients with a known intolerance of dapagliflozin
* Patients with high cardiovascular risk as specified by the most recent cardio-oncology guidelines.
* Patients with significant renal impairment (estimated glomerular filtration rate <45 mL/min/1.73 m2).
* Patients with a previous cancer diagnosis.
* Patients with known type 1 or 2 diabetes mellitus. We will not actively screen for diabetes. This is not done in clinical practice and there have been no issues.
* Patients with a contraindication to magnetic resonance imaging.
* Patients with prior exposure to anthracyclines.
* Patients who cannot read and understand English.
* Patients who are pregnant

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac energetics | From enrolment to the end of treatment at the end of approximately 22 weeks
  In vivo myocardial phosphocreatine/gamma-adenosine triphosphate (PCr/yATP) ratio by cardiac 31P cardiac magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Myocardial Ca2+ influx | From enrolment to the end of treatment at the end of approximately 22 weeks
  Myocardial Ca2+ influx assessed with manganese-enhanced magnetic resonance imaging (MEMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, MPhil, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baris VO, Dincsoy AB, Gedikli E, Zirh S, Muftuoglu S, Erdem A. Empagliflozin Significantly Prevents the Doxorubicin-induced Acute Cardiotoxicity via Non-antioxidant Pathways. Cardiovasc Toxicol. 2021 Sep;21(9):747-758. doi: 10.1007/s12012-021-09665-y. Epub 2021 Jun 5. PMID 34089496
- [Background] Maejima Y. SGLT2 Inhibitors Play a Salutary Role in Heart Failure via Modulation of the Mitochondrial Function. Front Cardiovasc Med. 2020 Jan 8;6:186. doi: 10.3389/fcvm.2019.00186. eCollection 2019. PMID 31970162
- [Background] Santos-Gallego CG, Requena-Ibanez JA, San Antonio R, Ishikawa K, Watanabe S, Picatoste B, Flores E, Garcia-Ropero A, Sanz J, Hajjar RJ, Fuster V, Badimon JJ. Empagliflozin Ameliorates Adverse Left Ventricular Remodeling in Nondiabetic Heart Failure by Enhancing Myocardial Energetics. J Am Coll Cardiol. 2019 Apr 23;73(15):1931-1944. doi: 10.1016/j.jacc.2019.01.056. PMID 30999996
- [Background] Selvaraj S, Fu Z, Jones P, Kwee LC, Windsor SL, Ilkayeva O, Newgard CB, Margulies KB, Husain M, Inzucchi SE, McGuire DK, Pitt B, Scirica BM, Lanfear DE, Nassif ME, Javaheri A, Mentz RJ, Kosiborod MN, Shah SH; DEFINE-HF Investigators. Metabolomic Profiling of the Effects of Dapagliflozin in Heart Failure With Reduced Ejection Fraction: DEFINE-HF. Circulation. 2022 Sep 13;146(11):808-818. doi: 10.1161/CIRCULATIONAHA.122.060402. Epub 2022 May 23. PMID 35603596
- [Background] Gaborit B, Ancel P, Abdullah AE, Maurice F, Abdesselam I, Calen A, Soghomonian A, Houssays M, Varlet I, Eisinger M, Lasbleiz A, Peiretti F, Bornet CE, Lefur Y, Pini L, Rapacchi S, Bernard M, Resseguier N, Darmon P, Kober F, Dutour A. Effect of empagliflozin on ectopic fat stores and myocardial energetics in type 2 diabetes: the EMPACEF study. Cardiovasc Diabetol. 2021 Mar 1;20(1):57. doi: 10.1186/s12933-021-01237-2. PMID 33648515
- [Background] Thirunavukarasu S, Jex N, Chowdhary A, Hassan IU, Straw S, Craven TP, Gorecka M, Broadbent D, Swoboda P, Witte KK, Cubbon RM, Xue H, Kellman P, Greenwood JP, Plein S, Levelt E. Empagliflozin Treatment Is Associated With Improvements in Cardiac Energetics and Function and Reductions in Myocardial Cellular Volume in Patients With Type 2 Diabetes. Diabetes. 2021 Dec;70(12):2810-2822. doi: 10.2337/db21-0270. Epub 2021 Oct 5. PMID 34610982
- [Background] Maslov MY, Chacko VP, Hirsch GA, Akki A, Leppo MK, Steenbergen C, Weiss RG. Reduced in vivo high-energy phosphates precede adriamycin-induced cardiac dysfunction. Am J Physiol Heart Circ Physiol. 2010 Aug;299(2):H332-7. doi: 10.1152/ajpheart.00727.2009. Epub 2010 May 21. PMID 20495142
- [Background] Govender J, Loos B, Marais E, Engelbrecht AM. Mitochondrial catastrophe during doxorubicin-induced cardiotoxicity: a review of the protective role of melatonin. J Pineal Res. 2014 Nov;57(4):367-80. doi: 10.1111/jpi.12176. Epub 2014 Oct 18. PMID 25230823
- [Background] Koleini N, Kardami E. Autophagy and mitophagy in the context of doxorubicin-induced cardiotoxicity. Oncotarget. 2017 Jul 11;8(28):46663-46680. doi: 10.18632/oncotarget.16944. PMID 28445146
- [Background] Goormaghtigh E, Chatelain P, Caspers J, Ruysschaert JM. Evidence of a complex between adriamycin derivatives and cardiolipin: possible role in cardiotoxicity. Biochem Pharmacol. 1980 Nov 1;29(21):3003-10. doi: 10.1016/0006-2952(80)90050-7. No abstract available. PMID 7458950
- [Background] Heck SL, Mecinaj A, Ree AH, Hoffmann P, Schulz-Menger J, Fagerland MW, Gravdehaug B, Rosjo H, Steine K, Geisler J, Gulati G, Omland T. Prevention of Cardiac Dysfunction During Adjuvant Breast Cancer Therapy (PRADA): Extended Follow-Up of a 2x2 Factorial, Randomized, Placebo-Controlled, Double-Blind Clinical Trial of Candesartan and Metoprolol. Circulation. 2021 Jun 22;143(25):2431-2440. doi: 10.1161/CIRCULATIONAHA.121.054698. Epub 2021 May 16. PMID 33993702
- [Background] Jones LW, Haykowsky MJ, Swartz JJ, Douglas PS, Mackey JR. Early breast cancer therapy and cardiovascular injury. J Am Coll Cardiol. 2007 Oct 9;50(15):1435-41. doi: 10.1016/j.jacc.2007.06.037. Epub 2007 Sep 24. PMID 17919562
- [Background] Lyon AR, Lopez-Fernandez T, Couch LS, Asteggiano R, Aznar MC, Bergler-Klein J, Boriani G, Cardinale D, Cordoba R, Cosyns B, Cutter DJ, de Azambuja E, de Boer RA, Dent SF, Farmakis D, Gevaert SA, Gorog DA, Herrmann J, Lenihan D, Moslehi J, Moura B, Salinger SS, Stephens R, Suter TM, Szmit S, Tamargo J, Thavendiranathan P, Tocchetti CG, van der Meer P, van der Pal HJH; ESC Scientific Document Group. 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS). Eur Heart J. 2022 Nov 1;43(41):4229-4361. doi: 10.1093/eurheartj/ehac244. No abstract available. PMID 36017568
- [Background] Felker GM, Thompson RE, Hare JM, Hruban RH, Clemetson DE, Howard DL, Baughman KL, Kasper EK. Underlying causes and long-term survival in patients with initially unexplained cardiomyopathy. N Engl J Med. 2000 Apr 13;342(15):1077-84. doi: 10.1056/NEJM200004133421502. PMID 10760308
- [Background] Zamorano JL, Lancellotti P, Rodriguez Munoz D, Aboyans V, Asteggiano R, Galderisi M, Habib G, Lenihan DJ, Lip GYH, Lyon AR, Lopez Fernandez T, Mohty D, Piepoli MF, Tamargo J, Torbicki A, Suter TM; ESC Scientific Document Group. 2016 ESC Position Paper on cancer treatments and cardiovascular toxicity developed under the auspices of the ESC Committee for Practice Guidelines: The Task Force for cancer treatments and cardiovascular toxicity of the European Society of Cardiology (ESC). Eur Heart J. 2016 Sep 21;37(36):2768-2801. doi: 10.1093/eurheartj/ehw211. Epub 2016 Aug 26. No abstract available. PMID 27567406